CLINICAL TRIAL: NCT01279343
Title: Cervical Foley Plus Vaginal Misoprostol Versus Vaginal Misoprostol for Cervical Ripening and Labor Induction: A Randomized Trial
Brief Title: Cervical Foley Plus Vaginal Misoprostol for Labor Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-1135-201107249
Record Dates: First submitted 2011-01-06; First posted 2011-01-19 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Induction of Labor
Keywords: labor induction; foley bulb; misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Foley Bulb plus Misoprostol (Experimental)
  Interventions: Device: Foley bulb
- Misoprostol (No Intervention)

INTERVENTIONS:
Device: Foley bulb — This is a randomized trial comparing foley bulb with the use of misoprostol versus use of misoprostol alone for cervical ripening and labor induction.
  Other Names: cytotec
  Arms: Foley Bulb plus Misoprostol

SUMMARY:
The purpose of this study is to compare the efficacy of the combination of the supracervical foley bulb and vaginal misoprostol to vaginal misoprostol alone for labor induction. We hypothesize that use of the foley bulb plus vaginal misoprostol will result in shorter induction to delivery time.

DETAILED DESCRIPTION:
More than 22% of all gravid women undergo induction of labor in the United States for various indications. Although there are several techniques and methods for induction of labor, the best agent and method still remains uncertain. To date, there has been no randomized trial comparing foley bulb plus vaginal misoprostol versus vaginal misoprostol alone. The combination of a mechanical device (foley bulb) and synthetic prostaglandin may have an additive or synergistic effect, resulting in greater degree of cervical ripening and shorter induction to delivery time (IDT). The addition of a synthetic prostaglandin to the foley bulb may also overcome the frequent observation of cervical dilation to 4cm by the foley bulb without effacement.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* vertex presentation
* unfavorable cervix(Bishop's score less than or equal to 6)
* greater than 24 weeks gestation

Exclusion Criteria:

* fetal malpresentation
* multifetal gestation
* spontaneous labor
* more than 5 uterine contractions in 10 minutes
* contraindication to prostaglandins
* non-reassuring fetal heart rate tracing
* intrauterine growth restriction
* anomalous fetus
* fetal demise
* previous cesarean delivery or other significant uterine surgery

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine F Carbone, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Result] Carbone JF, Tuuli MG, Fogertey PJ, Roehl KA, Macones GA. Combination of Foley bulb and vaginal misoprostol compared with vaginal misoprostol alone for cervical ripening and labor induction: a randomized controlled trial. Obstet Gynecol. 2013 Feb;121(2 Pt 1):247-252. doi: 10.1097/AOG.0b013e31827e5dca. PMID 23303106
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

RESULTS

PARTICIPANT FLOW:
Groups:
- Foley Bulb Plus Misoprostol: In the combination arm participants received vaginal misoprostol at 25 micrograms every 4 hours. The foley bulb was also inserted in these participants.
- Misoprostol: The participants in this arm received misoprostol 25 micrograms every 4 hours.
Period: Overall Study
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Started | 59 | 64
Completed | 57 | 58
Not Completed | 2 | 6
Not completed — Did not receive treatment | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol | Total
Number analyzed (Participants) | 56 | 61 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (7.2) | 24.2 (5.5) | NA (NA) — Data not available because PI has left the institution,additional result information is not available.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 61 | 117
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 40 | 74
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 56 | 61 | 117
Maternal weight [Mean (Standard Deviation); unit: kg] | 89.6 (20.3) | 90.6 (24.9) | NA (NA) — Data not available because PI has left the institution,additional result information is not available.
Indication for labor inductions [Count of Participants; unit: Participants]
  Postdates | 24 | 26 | 50
  Preeclampsia | 7 | 8 | 15
  Chronic Hypertension | 4 | 4 | 8
  Pregnancy induced hyptertension | 2 | 2 | 4
  Pregestational diabetes | 2 | 4 | 6
  Gestational diabetes | 3 | 2 | 5
  Oligohydramnios | 2 | 1 | 3
  Elective | 6 | 8 | 14
  Other | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Labor Induction to Vaginal Delivery
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
hour | 15.3 (6.5) | 18.3 (8.7)
Statistical Analysis 1: Comparison: Foley Bulb Plus Misoprostol vs Misoprostol; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-5.9 to -0.3]

2. Secondary Outcome: Successful Number of Vaginal and Cesarean Deliveries
Description: To compare the number of vaginal deliveries to failed inductions requiring cesarean deliveries.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
Participants
  Vaginal delivery | 41 | 45
  Cesarean delivery | 15 | 16
Statistical Analysis 1: Comparison: Foley Bulb Plus Misoprostol vs Misoprostol; Comparison of vaginal delivery between groups; Test type: Superiority; p = 0.96, Chi-squared; Risk Ratio (RR) = 0.99, 95% CI 2-sided [.80 to 1.23]
Statistical Analysis 2: Comparison: Foley Bulb Plus Misoprostol vs Misoprostol; Cesarean deliveries were compared between the groups; Test type: Superiority; p = 0.90, Chi-squared; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.57 to 1.90]

3. Secondary Outcome: Number of Participants Experiencing Tachysystole With Deceleration
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
Participants | 10 | 12

4. Secondary Outcome: Number of Participants With Post-partum Hemorrhage
Time Frame: 96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
Participants | 2 | 5

5. Secondary Outcome: Chorioamnionitis
Time Frame: 96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
Participants | 5 | 7

6. Secondary Outcome: Neonatal APGAR Scores
Description: APGAR scores will be recorded at 1 and 5 minutes after birth. In the test, five things are used to check a baby's health. Each is scored on a scale of 0 to 2, with 2 being the best score:
  Appearance (skin color) Pulse (heart rate) Grimace response (reflexes) Activity (muscle tone) Respiration (breathing rate and effort)
Time Frame: 5 minutes
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
score on a scale
  1 minute apgar scord | 8 [2 to 9] | 8 [2 to 9]
  5 minute apgar score | 9 [1 to 9] | 9 [7 to 9]

7. Secondary Outcome: NICU Admission
Time Frame: 96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
Participants | 0 | 2

8. Secondary Outcome: Time to Complete Cervical Dilation
Description: We will record the start time of induction until the patient's cervix is 10cm dilated
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
hour | 13.7 (5.9) | 17.1 (8.7)

9. Secondary Outcome: Delivery Within 24 Hours
Time Frame: Delivery within 24 hours of induction
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
Participants | 49 | 46

10. Secondary Outcome: Admission to NICU or Special Care Nursery
Time Frame: birth to 96 hours of age
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Number analyzed (Participants) | 56 | 61
Participants | 8 | 11

ADVERSE EVENTS:
Description: PI has left the institution and no adverse event information is available for this study.
Arm/Group | Foley Bulb Plus Misoprostol | Misoprostol
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No